CLINICAL TRIAL: NCT02234661
Title: Expanding the Cycle of Opportunity: Simultaneously Educating Parents and Children in Head Start
Acronym: CAPFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lindsay Chase-Lansdale, Frances Willard Professor of Human Development and Social Policy Associate Provost for Faculty, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ACF Grant # 90YR0073
Record Dates: First submitted 2014-08-07; First posted 2014-09-09 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Children; Parents
Keywords: Low income; Education; Poverty; Children; Parents; Head Start

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CareerAdvance® (Experimental): CareerAdvance® provides education, career coaching, and soft-skills training for parents while their children attend Head Start programs.
  Interventions: Behavioral: CareerAdvance®
- Control Standard of CAP (No Intervention): Control participants access to CAP array of service

INTERVENTIONS:
Behavioral: CareerAdvance® — CareerAdvance® is a dual-generation program providing education, career coaching, and soft-skills training for parents while their children attend CAP Tulsa's Head Start programs.
  Arms: CareerAdvance®

SUMMARY:
The CAP Family Advancement Study (CAP FAST) is a randomized control trial of CareerAdvance®, a dual-generation program providing education, career coaching, and soft-skills training for parents while their children attend CAP Tulsa's Head Start programs.

DETAILED DESCRIPTION:
Randomization will take place with all applicants who have agreed to the study and are selected to participate in CareerAdvance®. Two-thirds of participants will be selected for the treatment group and will be able to enroll in CareerAdvance® immediately. The other one-third of the participants will be assigned to the control group and will not be able to enroll in CareerAdvance® for two years. Those who are selected for the control group will have access to CAP Tulsa's rich array of service outside of CareerAdvance®, including high quality early childhood education. The randomization process is introduced to parents during CareerAdvance® information sessions, and consent for the randomization process is required in order to apply to CareerAdvance®.

ELIGIBILITY:
Inclusion Criteria:

* Families whose children attend CAP Tulsa's Early Head Start and Head Start programs, and whose parents have applied to CareerAdvance®.

Exclusion Criteria:

* Participants who have not applied to CareerAdvance®..

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2014-06; Primary Completion 2020-06 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Parent's educational achievement | 16 months
  Defined education course credit attainment

CONTACTS AND LOCATIONS:
Overall Officials: P. Lindsay Chase-Lansdale, PhD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Evanston, Illinois
  - Oklahoma State University, Tulsa, Oklahoma
  - Community Action Project of Tulsa County, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study description and publications via website — https://sites.northwestern.edu/nu2gen/sample-page/current-studies/immigrant-families/